CLINICAL TRIAL: NCT05211362
Title: Sticky Bone and Repeated Injectable PRF Application in Management of Periodontal Intrabony Defects (Randomized Clinical Trial)
Brief Title: Sticky Bone and Repeated Injectable PRF (iPRF) Application in Management of Periodontal Intrabony Defects
Acronym: IPRF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mahmoud eldestawy, associate professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 748/2757
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Sticky Bone; iPRF; Periodontal Defect
Keywords: iPRF; sticky bone graft
MeSH Terms: interventions — Bone Substitutes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sticky Bone and Repeated Injectable PRF (iPRF) (Experimental): The surgical treatment phase was initiated only if the subjects had a full-mouth dental plaque score of less than one and a test site plaque score of 0. Following mucoperiosteal flap reflection for one tooth on either side of the defect, all granulation tissue was removed from the defects by means of Gracey 7/8 metal curettes, and root surfaces were scaled and planed using hand and ultrasonic instruments, then the defect was filled with xenograft mixed with IPRF, Finally, the flap was replaced and closed with crossed horizontal and vertical internal mattress sutures.
  Interventions: Biological: Sticky Bone and Repeated Injectable PRF (iPRF)
- bone substitute (Active Comparator): The surgical treatment phase was initiated only if the subjects had a full-mouth dental plaque score of less than one and a test site plaque score of 0. Following mucoperiosteal flap reflection for one tooth on either side of the defect, all granulation tissue was removed from the defects by means of Gracey 7/8 metal curettes, and root surfaces were scaled and planed using hand and ultrasonic instruments, bone graft substitute was heavily condensed into the intra bony defects. The flap was replaced and closed with crossed horizontal and vertical internal mattress sutures.
  Interventions: Biological: bone substitute

INTERVENTIONS:
Biological: Sticky Bone and Repeated Injectable PRF (iPRF) — The surgical treatment phase was initiated only if the subjects had a full-mouth dental plaque score of less than one and a test site plaque score of 0. Following mucoperiosteal flap reflection for one tooth on either side of the defect, all granulation tissue was removed from the defects by means of Gracey 7/8 metal curettes, and root surfaces were scaled and planed using hand and ultrasonic instruments, then the defect was filled with xenograft mixed with IPRF, Finally, the flap was replaced and closed with crossed horizontal and vertical internal mattress sutures.
  Arms: Sticky Bone and Repeated Injectable PRF (iPRF)
Biological: bone substitute — The surgical treatment phase was initiated only if the subjects had a full-mouth dental plaque score of less than one and a test site plaque score of 0. Following mucoperiosteal flap reflection for one tooth on either side of the defect, all granulation tissue was removed from the defects by means of Gracey 7/8 metal curettes, and root surfaces were scaled and planed using hand and ultrasonic instruments, bone graft substitute was heavily condensed into the intra bony defects. The flap was replaced and closed with crossed horizontal and vertical internal mattress sutures.
  Arms: bone substitute

SUMMARY:
One of the main objectives of periodontal therapy is the regeneration of the tooth's supporting periodontal tissue to its original levels. The healing after non-surgical and conventional surgical methods is histologically characterized by a long junctional epithelium along the root surfaces. Therefore, reconstructive techniques are required. Although complete periodontal regeneration is unpredictable with any regenerative therapy currently used, so the objective of our trial is to get complete periodontal regeneration by using Sticky Bone and Repeated Injectable PRF (iPRF) in Management of Periodontal Intrabony Defects.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases which could influence the outcome of therapy.
* Good compliance with plaque control instructions following initial therapy.
* Teeth involved were all vital with no mobility.
* Each subject contributed a single predominately 2 or 3-wall intrabony interproximal defect around premolar or molar teeth without furcation involvement
* Selected intrabony defects (IBD) measured from the alveolar crest to the defect base in diagnostic periapical radiographs of ≥ 3 mm, the width of ≥ 3 mm at its most coronal part, with no cratering that involve both mesial and distal surfaces of adjacent teeth.
* Selected probing depth (PD) ≥ 6 mm and clinical attachment loss (CAL) ≥ 4 mm at the site of intraosseous defects four weeks following initial cause-related therapy.
* Availability for the follow-up and maintenance program; 8) absence of periodontal treatment during the previous year.

Exclusion Criteria:

• Pregnant females.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-16 (Estimated); Primary Completion 2022-08-25 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
change in clinical attachment level | baseline, 3, and 6 months
  change in clinical attachment level

SECONDARY OUTCOMES:
change in interseptal bone width | baseline, 3, and 6 months
  change in interseptal bone width

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud eldestawy, associted profissor, Principal Investigator — al azhar universty
Locations (1):
- Mah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol